CLINICAL TRIAL: NCT02034240
Title: Secretion of Neutrophil Gelatinase Associated Lipocalin in Septic Patients and the Development of Acute Kidney Injury
Brief Title: Neutrophil Gelatinase Associated Lipocalin (NGAL) in Urine: Can This Prove to be a Biomarker for Acute Kidney Injury in Patients With Sepsis?
Status: Completed | Type: Observational
Sponsor: Sygehus Lillebaelt (Other)
Collaborators: Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Claes Falkenberg Elvander, Medical Doctor, Sygehus Lillebaelt
Other Study IDs: DNVK:1305 385
Record Dates: First submitted 2014-01-07; First posted 2014-01-13 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Severe Sepsis; Septic Shock; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Patient Registry: Yes
Target Follow-Up Duration: 5 Weeks
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with severe infection and sepsis are in high risk of hypo perfusion and therefore organ affection. Temporary or permanent kidney failure is a common complication in these patients. Today's golden standard for kidney failure detection is creatinine levels rising and / or oliguria. The investigators hypothesize that an even more sensitive biomarker; neutrophil gelatinase associated lipocalin(NGAL) in urine can predict kidney injury before creatinine levels rise. In recent studies NGAL in urine seem to be a sensitive biomarker in these patient to predict kidney injury, but the time factor for sampling optimally is not known. In this pilot study the investigators sample the urine at admission within the first hour of hospitalization to investigate if NGAL can be used as a predictor in an emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis
* Septic shock
* Patients must not be able to give consent

Exclusion Criteria:

* Underaged (18 years )
* known kidney injury
* Fully alert patients that can give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with no prior record of kidney failure
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Development of Acute Kidney Failure | During hospitalization, anticipated approximately 5 weeks

SECONDARY OUTCOMES:
Levels of NGAL in patients with kidney failure compared to creatinine | During hospitalization, anticipated approximately 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jannie Bisgaard Stæhr, PhD, M.D, Study Chair — Odense University Hospital; Claes Falkenberg Elvander, M.D, Study Director — Kolding Sygehus; Srishamanthi Sriskandarajah, M.D, Principal Investigator — Kolding Sygehus
Locations (1):
- Faelles Akut Modtagelse, Kolding Sygehus, Kolding, Denmark